CLINICAL TRIAL: NCT02423694
Title: Effectiveness and Safety of Electro-acupuncture for Mild-to-moderate Perimenopausal Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Fu Wenbin, Professor, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012BAI24B01
Record Dates: First submitted 2015-04-11; First posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Perimenopause; Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Electroacupuncture (Experimental): Baihui, Yintang, Guanyuan(dual), Zigong(dual), Sanyinjiao(dual), Hegu(dual), Taichong(dual).
  Insert needles to the acupoints mentioned above after sterilized.Needle handles of Baihui and Yintang are connected with the electroacupuncture instrument wire. And needle handles of bilateral Zigong are conneted with the electroacupunture instrument wire. And needle handles of bilateral Tianshu are connected with the electroacupunture instrument wire. Density wave, frequency of 10/50Hz and current intensity is 0.5~1.0 mA for 30 minutes. 3 times per week. Each treatment interval of more than 24 hours, continuous treatment for 12 weeks.
  Interventions: Device: electro-acupuncture
- escitalopram oxalate tablets (Active Comparator): 0.5 hour after breakfast oral taking 10mg escitalopram oxalate tablets, continuous treatment for 12 weeks.
  Interventions: Drug: escitalopram oxalate tablets

INTERVENTIONS:
Device: electro-acupuncture — 8 acupoint: Guanyuan, Zigong (bilateral), Tianshu(bilateral), Sanyinjiao(bilateral), Hegu(bilateral), Taichong(bilateral), Baihui, Yintang.
  Every patient is supposed to have 36 times acupuncture treatment. 30 minutes per time. Baihui, Yintang, Zigong (bilateral), Tianshu (bilateral) are applied with electro-acupuncture device with dilatational wave, current frequency: 10/50Hz, intensity: 0.5~1.0 mA
  Arms: Electroacupuncture
Drug: escitalopram oxalate tablets — escitalopram oxalate tablet, once a day, 0.5 hour after breakfast, oral taken, 10mg, for 12 weeks
  Arms: escitalopram oxalate tablets

SUMMARY:
Main objective: to compare the effects of electro-acupuncture and escitalopram oxalate tablets on mild-to-moderate perimenopausal depression, and to evaluate the safety of electroacupuncture stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Conforms to the diagnosis standard of STRAW-10 for perimenopause, conforms to the diagnosis standard of The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) for depression, and conforms to the diagnosis standard of The International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) F32.0(mild depression) or F32.1(moderate depression);
* Fisrt attack during perimenopausal period;
* HAMD-17 score >7 and <23;
* Age ≥45 to ≤55;
* No hormone replacement therapy (HRT) or no antidepressant 3 months before into the group;
* Sign the consent consent, volunteered for this study

Exclusion Criteria:

* Fail to rule out the possibility of suicide in depression factor of The Symptom Checklist (SCL-90);
* Application of estrogen, progesterone, selective serotonin reuptake inhibitors (SSRIs), soybean isoflavone, vitamin E or black cohosh in recent 4 weeks;
* Allergic to citalopram or escitalopram tablets;
* Taken the non selective, irreversible inhibitor of monoamine oxidase (MAOIs) in recent 2 weeks;
* Taken linezolid, pimozide, tryptophane,tramadol, triptans or other drugs that may cause drug adverse reactions in recent 2 weeks;
* Patient with prolongation of the QT interval or congenital long QT syndrome
* Taken herbs or products that contain isatin, pilose antler, hawthorn, fleeceflower root, common St.John's wort herb, hypericin;
* Ovarian dropsy or hysteromyoma with more than 4cm diameter, oophorectomy, or hysterectomy;
* Mandatory indications of hormonotherapy, such as surgery-induced menopause or osteoporosis;
* Patient with history of radiotherapy or chemotherapy, or undergoing radiotherapy or chemotherapy;
* Vaginal bleeding of undetermined origin;
* Patient with coagulation disorders, or taking anticoagulants such as Warfarin, or heparin;
* Patient with skin diseases, such as eczema,or psoriasis;
* Serious hepatic insufficiency or serious renal inadequacy;
* Uncontrolled hypertension, diabetes, or thyroid disease;
* Diabetic neuropathy, or malignant tumor;
* Pregnancy intention, in pregnancy or lactation;
* Regular use of sedative and anti anxiety drugs;
* The long-term smoking and/or drinking;
* Having Pacemaker or artificial joint；
* Electrolyte is disorder, serious heart disease or other potential life-threatening disease patients;
* Compliance may be poor or fear of acupuncture.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in scores of the 17-item Hamilton depression rating scale (HAMD-17) | 0 week, 4th week, 8th week, 12th week, 16th week and 24th week

SECONDARY OUTCOMES:
Change from Baseline in scores of the Menopause-Specific Quality of Life questionnaire (MENQOL) | 0 week, 4th week, 8th week, 12th week, 16th week, 20th week and 24th week
Change from Baseline in level of estradiol (E2), | 0 week, 12th week
Change from Baseline in level of follicle-stimulating hormone (FSH) | 0 week, 12th week
Change from baseline in level of Luteinizing hormone (LH) | 0 week, 12th week
Change from baseline in level of FSH/LH | 0 week, 12th week

OTHER OUTCOMES:
safety of electro-acupuncture as measured by safety and acceptability questionnaires | 0 week, 4th week, 8th week, and 12th week
  safety and acceptability
safety of escitalopram as measured by Asberg Rating Scale for Side Effect (SERS) | 0 week, 4th week, 8th week, and 12the week
  Asberg Rating Scale for Side Effect (SERS)
safety of escitalopram as measured by liver functure test | 0 week, 4th week, 8th week, and 12the week
  ALT, aspartate transminase (AST), and TBIL
safety of escitalopram as measured by kidney functure test | 0 week, 4th week, 8th week, and 12the week
  Cr, BUN
safety of both groups before treatment as measured by EKG | 0 week
  EKG
safety of both groups before treatment as meausred by blood regular test | 0 week
  Blood regular test
safety of both groups before treatment as measured by urine regular test | 0 week
  Urine regular test

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Fu, MD, Study Chair — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Li S, Li ZF, Wu Q, Guo XC, Xu ZH, Li XB, Chen R, Zhou DY, Wang C, Duan Q, Sun J, Luo D, Li MY, Wang JL, Xie H, Xuan LH, Su SY, Huang DM, Liu ZS, Fu WB. A Multicenter, Randomized, Controlled Trial of Electroacupuncture for Perimenopause Women with Mild-Moderate Depression. Biomed Res Int. 2018 May 29;2018:5351210. doi: 10.1155/2018/5351210. eCollection 2018. PMID 30003102